CLINICAL TRIAL: NCT07055035
Title: Clinical Study on the Application of Two-dimensional Speckle Tracking Imaging to Evaluate the Atrial Synchrony of Bachmann Bundle Pacing in Patients With Sick Sinus Syndrome
Brief Title: Atrial Synchrony Evaluation of Bachmann Bundle Pacing in Sick Sinus Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyan City Renmin Hospital (Other Government)
Responsible Party: Principal Investigator, You Wu, Principal Investigator, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025126x
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Sick Sinus Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bachmann Bundle Pacing (BBP) Group (Experimental): Patients were randomized to receive a permanent pacemaker with the atrial lead placed in the Bachmann bundle region. They were followed up at 1 month and 3 months post-procedure.
  Interventions: Device: Bachmann Bundle Pacing
- Right Atrial Appendage (RAA) Pacing Group (Active Comparator): Patients were randomized to receive a permanent pacemaker with the atrial lead placed in the conventional right atrial appendage. They were followed up at 1 month and 3 months post-procedure.
  Interventions: Device: Right Atrial Appendage Pacing

INTERVENTIONS:
Device: Bachmann Bundle Pacing — Implantation of a permanent pacemaker system. The atrial lead (Medtronic 3830 active electrode) is surgically positioned and fixed in the Bachmann bundle region, located at the angle between the superior vena cava and the atrium in the mid-posterior position of the high atrial septum. Successful placement is confirmed by achieving a P-wave width shortening of at least 30ms compared to the preoperative P-wave. The ventricular lead is positioned in the mid-to-lower portion of the ventricular septum. Pacing parameters are measured and confirmed to be good.
  Arms: Bachmann Bundle Pacing (BBP) Group
Device: Right Atrial Appendage Pacing — Implantation of a permanent pacemaker system using the conventional technique. The atrial active electrode is surgically positioned and fixed in the right atrial appendage. The ventricular lead is placed in the mid-to-lower portion of the ventricular septum. Pacing parameters (sensing > 2.0mV; impedance between 300 to 1000Ω; threshold < 1.5mV) are confirmed to be good.
  Arms: Right Atrial Appendage (RAA) Pacing Group

SUMMARY:
This is a prospective, randomized study to compare the effects of Bachmann bundle pacing (BBP) versus conventional right atrial appendage (RAA) pacing on atrial electromechanical synchrony in patients with sick sinus syndrome (SSS). The study utilizes two-dimensional speckle tracking imaging (2D-STI) to assess improvements in cardiac function and synchrony, aiming to determine a more optimal pacing site for SSS patients.

DETAILED DESCRIPTION:
Sick sinus syndrome (SSS) is a common indication for permanent pacemaker implantation. Conventional right atrial appendage (RAA) pacing, however, is non-physiological and may lead to atrial conduction delays, atrial remodeling, and an increased risk of atrial fibrillation. Bachmann bundle pacing (BBP) is emerging as a more physiological pacing strategy that may correct atrial conduction delays and improve electromechanical synchronization. This study prospectively enrolled and randomized 72 patients with SSS to receive either BBP or RAA pacing. The primary objective is to evaluate the differences in atrial synchrony, cardiac function, and pacing parameters between the two groups at baseline, 1-month, and 3-month follow-ups, using electrocardiography and two-dimensional speckle tracking imaging (2D-STI). The study aims to provide evidence for BBP as a superior treatment option for improving long-term outcomes in SSS patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for sick sinus syndrome (e.g., persistent sinus bradycardia <50 bpm, sinus arrest, sinoatrial block, or tachy-brady syndrome).
* Age between 30 and 90 years.
* Has not taken any other antiarrhythmic drugs within one month prior to enrollment.
* Has not participated in any other related clinical trials.
* Voluntarily signs the informed consent form.

Exclusion Criteria:

* Patients with severe primary diseases causing unstable vital signs (e.g., severe circulatory, digestive, or neurological system diseases).
* Patients with a history of recurrent syncope, Adams-Stokes syndrome, severe bradycardia (lowest sinus rhythm <30 bpm), or long RR interval >3s.
* Pregnant or lactating women.
* Patients with mental illness.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Inter-atrial Electromechanical Delay (Inter AEMD) | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured by two-dimensional speckle tracking imaging (2D-STI) as the time difference between the onset of the P-wave on the electrocardiogram (ECG) and the peak longitudinal strain of the lateral walls of the right and left atria. A smaller value indicates better inter-atrial synchrony.
Change in Intra-atrial Mechanical Delay (IAMD) | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured by 2D-STI as the standard deviation of the time-to-peak longitudinal strain of six segments of the left atrium. A smaller value indicates better intra-atrial synchrony.
Change in Intra-right Atrial Electromechanical Delay (Intra-right AEMD) | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured by 2D-STI as the time difference between the earliest and latest peak longitudinal strain within the right atrium segments.

SECONDARY OUTCOMES:
Change in P-wave Duration (PWD) and Morphology | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured from the 12-lead surface ECG, including P-wave duration (P-AT, P-Am) and P-wave axis (P-aI, P-aL).
Change in QRS Duration and Axis | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured from the 12-lead surface ECG.
Change in Left Atrial (LA) and Right Atrial (RA) Dimensions | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured by standard 2D echocardiography.
Change in Left Ventricular End-Systolic Diameter (LVESD) and End-Diastolic Diameter (LVEDD) | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Measured by standard 2D echocardiography.
Change in Left Atrial Strain Parameters | Baseline, 1 Month Post-procedure, 3 Months Post-procedure
  Includes left atrial reservoir strain (LASr), conduit strain (LAScd), and contraction strain (LASct), measured by 2D-STI.
Recurrence of Atrial Arrhythmia | Up to 1 year
  Number of patients experiencing newly developed or recurrent atrial fibrillation or atrial tachycardia.
Change in Atrial Pacing Threshold | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: millivolts (mV).
Change in Atrial Sensing (P-wave amplitude) | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: millivolts (mV).
Change in Atrial Pacing Impedance | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: Ohms (Ω).
Change in Ventricular Pacing Threshold | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: millivolts (mV).
Change in Ventricular Sensing (R-wave amplitude) | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: millivolts (mV).
Change in Ventricular Pacing Impedance | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: Ohms (Ω).
Percentage of Ventricular Pacing | 1 Month Post-procedure, 3 Months Post-procedure
  Measured via pacemaker programmer interrogation. Unit: Percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Wu, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Shiyan, Hubei, China